CLINICAL TRIAL: NCT06895291
Title: Whole Body MRI in Oncology
Acronym: ONCO-MRI
Status: Recruiting | Type: Observational
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRST100.61
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Lymphoma; Advanced Prostate Cancer; Advanced Breast Cancer; Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma; Multiple Myeloma
Keywords: Monoclonal Gammopathy of Undetermined Significance; Smoldering multiple myeloma; Multiple myeloma; Advanced Breast Cancer; Advanced Prostate Cancer; Lymphoma; Whole Body-Magnetic Resonance Imaging
MeSH Terms: conditions — Lymphoma; Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients affected by Monoclonal plasma cell disorders: Monoclonal Gammopathy of Undetermined Significance (MGUS), Smoldering Multiple Myeloma (SMM), Multiple Myeloma (MM).
  Interventions: Diagnostic Test: Whole Body-Magnetic Resonance Imaging (WB-MRI)
- Patients affected by advanced prostate cancer (APC) or advanced breast cancer (ABC): Patients affected by advanced prostate (APC) or breast cancer (ABC) with high suspicious of metastasis particularly in case of diagnostic doubt in other imaging methods (Computed tomography (CT), Positron Emission Computed Tomography (PET/CT), Bone Scintigraphy (BS)).
  Interventions: Diagnostic Test: Whole Body-Magnetic Resonance Imaging (WB-MRI)
- Patients affected by Lymphomas.: Patients affected by Lymphomas.
  Interventions: Diagnostic Test: Whole Body-Magnetic Resonance Imaging (WB-MRI)

INTERVENTIONS:
Diagnostic Test: Whole Body-Magnetic Resonance Imaging (WB-MRI) — This is a non-pharmacological, observational, prospective, study. Each patient will undergo quantitative WB-MRI as per clinical routine. WB-MRI may be performed:
  * at staging
  * at follow-up Disease progression is defined by clinicians taking into account all imaging modalities and clinicolaboratorial data available for the patients.

SUMMARY:
Multicenter, observational, prospective, study. All patients will be treated and monitored according to the local clinical practice. No additional procedures/patient visits in comparison with the usual clinical practice are planned for the study.

DETAILED DESCRIPTION:
Whole Body-Magnetic Resonance Imaging (WB-MRI) is a radiation-free and, usually, contrast administration-free imaging method for detecting bone and soft tissue pathology. It's part of the "next generation imaging techniques" combining high quality morphological images with "functional" information on diffusivity of water molecules through diffusion- weighted sequences (DWI).

Nowadays WB-MRI has been introduced in several guidelines in oncological settings, in particular for staging and relapse in patients affected by monoclonal plasma cell disorders, screening in patients with cancer predisposition syndromes (Li fraumeni syndrome, hereditary paraganglioma / pheochromocytoma syndrome, neurofibromatosis) and staging and follow-up of cancer patients affected by predominant bone metastatic pattern, particularly advanced prostate cancer and breast cancer.

The current limit on the diffusion of the technique is that it is not widely available as it requires an optimal set up of both the machine with specific sequences and the acquisition protocol, as well as dedicated, trained staff.

DWI is emerging as a core sequence of WB-MRI protocols for disease assessment because of its sensitiveness to tissue cellularity and cell viability offering excellent lesion-to-background contrast and quantification of the degree of water motion by calculation of the apparent diffusion coefficient (ADC); changes in ADC can reflect variations in cellularity. Fat-Fraction (FF) is another emerging sequence for tissue characterization that quantifies the relative amount of fat. A better investigation of these novel sequences can maximize sensitivity and specificity in order to improve our understanding of diseases assessment.

The aim of this observational study is to evaluate whether WB-MRI allows an improvement in identification of site of tumour disease or earlier progression in comparison to other methodologies that are nowadays the standard of care due to their widespread availability in hospitals and quicker execution, particularly Bone Scintigraphy (BS) Computed Tomography (CT), Positron Emission Tomography/Computed Tomography (PET/CT) .

ELIGIBILITY:
Inclusion Criteria:

* Patients candidate to WB-MRI according to clinical practice belonging to the study groups listed above.
* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged ≥ 18 years.
* Life expectancy greater than 3 months.

Exclusion Criteria:

* Patients with MRI-unsafe prostheses and devices.
* Patients whose tests are of suboptimal quality, or whose test has been suspended, or is incomplete.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The following patients groups will be prospectively enrolled:
  * Patients affected by Monoclonal plasma cell disorders (monoclonal gammopathy of undertermined significance-MGUS, Smoldering multiple myeloma- SMM, Multiple myeloma-MM).
  * Patients affected by advanced prostate (APC) or breast cancer (ABC) with high suspicious of metastasis particularly in case of diagnostic doubt in other imaging methods (CT, PET/CT, BS).
  * Patients affected by Lymphomas.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate whether WB-MRI allows a better evaluation of bone marrow involvement and/or soft tissue lesions in different kind of pathologies in comparison to other standard imaging modalities. | 36 months
  To evaluate the accuracy of WB-MRI in terms of:
  Myeloma: pattern of bone marrow or soft tissues involvement (Negative /Micronodular/ diffuse/focal/ focal on diffuse/ extra and perimedullary disease)
To evaluate whether WB-MRI allows a better evaluation of bone marrow involvement and/or soft tissue lesions in different kind of pathologies in comparison to other standard imaging modalities. | 36 months
  To evaluate the accuracy of WB-MRI in terms of:
  -Metastatic breast cancer an Metastatic prostate cancer: Number of lesions for oligometastatic patients or diffuse pattern for diffuse bone marrow involvement
To evaluate whether WB-MRI allows a better evaluation of bone marrow involvement and/or soft tissue lesions in different kind of pathologies in comparison to other standard imaging modalities. | 36 months
  To evaluate the accuracy of WB-MRI in terms of:
  -Lymphoma:number of lesions will be assessed.
To evaluate whether WB-MRI allows a better evaluation of bone marrow involvement and/or soft tissue lesions in different kind of pathologies in comparison to other standard imaging modalities. | 36 months
  To evaluate the accuracy of WB-MRI in terms of:
  -Lymphoma:diameters of lesions will be assessed.
To evaluate whether WB-MRI allows earlier identification of disease progression in comparison to other standard methodologies and to assess different patterns of response, stable disease, and progression that can be observed on WB-MRI. | 36 months
  Pattern of response/progression will be determined in terms of:
  -Myeloma:Myeloma Response Assessment and Diagnosis System (MY-RADS) criteria will be applied on WB-MRI whereas n.of lesions and lesion uptake Standardized Uptake Value (SUV) variations will be used to evaluate PET-CT response.
To evaluate whether WB-MRI allows earlier identification of disease progression in comparison to other standard methodologies and to assess different patterns of response, stable disease, and progression that can be observed on WB-MRI. | 36 months
  Pattern of response/progression will be determined in terms of:
  -Metastatic prostate cancer and Metastatic breast cancer: soft tissue response and progression on CT will be assessed according to RECIST 1.1guidelines. Definitions of complete and partial response or progression for bone lesions on CT and/or BS have been adopted from MD Anderson (MDA) criteria for ABC and from Prostate Cancer Working Group3 (PCWG3) for APC.
To evaluate whether WB-MRI allows earlier identification of disease progression in comparison to other standard methodologies and to assess different patterns of response, stable disease, and progression that can be observed on WB-MRI. | 36 months
  Pattern of response/progression will be determined in terms of:
  -Lymphoma:for Contrast-Enhanced Computed Tomography (CE-CT) and PET-CT Lugano criteria or Lymphoma Response to Immunomodulatory Therapy Criteria criteria will be used
To evaluate whether WB-MRI allows earlier identification of disease progression in comparison to other standard methodologies and to assess different patterns of response, stable disease, and progression that can be observed on WB-MRI. | 36 months
  Pattern of response/progression will be determined in terms of:
  -Lymphoma:for the diameter evaluation of max 5 lymphnodes or lesion integrated with apparent diffusion coefficient (ADC) evaluation will be applied on WB-MRI.
To evaluate how WB-MRI, added to other imaging modalities, alters decision making and management of patients. | 36 months
  The number of times a patient treatment's course was changed by clinicians after evidences provided by WB-MRI investigations as per clinical routine.

SECONDARY OUTCOMES:
Identification of imaging biomarkers for precise disease differentiation or for response prediction. | 36 months
  We will evaluate the discriminating performance of imaging features for differentiating between smouldering multiple myeloma and multiple myeloma.
Identification of imaging biomarkers for precise disease differentiation or for response prediction. | 36 months
  We will assess the discriminating performance of imaging features for differentiating between invasive lobular carcinoma and invasive ductal carcinoma.
Identification of imaging biomarkers for precise disease differentiation or for response prediction. | 36 months
  We will examine the discriminating performance of imaging features for distinguishing between the heterogeneous histotype characteristics of lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Rossi, Principal Investigator — IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l.
Locations (3):
- Italy (3):
  - IRCCS - Azienda Ospedaliero-Universitaria di Bologna - Policlinico di S. Orsola, Bologna, BO
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l., Meldola, FC
  - IRCCS Istituto Europeo di Oncologia S.r.l., Milan, MI

IPD SHARING:
Plan to Share IPD: No